CLINICAL TRIAL: NCT04429074
Title: Registrar Performance in Laparoscopic Distal Pancreatectomy and Its Effect on Postoperative Outcomes
Brief Title: Registrar Performances in MIDP
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0348
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Minimally Invasive Distal Pancreatectomy
Keywords: Benign or borderline pathology (non-pancreatic cancer); laparoscopy; registrar; postoperative outcomes; pancreatectomy; surgery; pancreas

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Registrar): Group 1 (Registrar): Patients who underwent minimally invasive distale pancreatectomy for benign or borderline pathology operated on by a registrar (young specialist surgeon)
  Interventions: Procedure: Minimally invasive distal pancreatectomy
- Group 2 (Consultant): Group 2 (Consultant): Patients who underwent minimally invasive distale pancreatectomy for benign or borderline pathology operated on by a consultant (expert)
  Interventions: Procedure: Minimally invasive distal pancreatectomy

INTERVENTIONS:
Procedure: Minimally invasive distal pancreatectomy — Minimally invasive distal pancreatectomy

SUMMARY:
This study aimed to determine whether registrar involvement in minimally invasive distal pancreatectomy (MIDP) was associated with adverse outcomes.

DETAILED DESCRIPTION:
From January 2009 to March 2020, data of all consecutive patients requiring distal pancreatectomy in our public tertiary hospital were prospectively collected and retrospectively analyzed.

Registrars were progressively involved for MIDP since 2009 and their experience was: < 5 open pancreatic resections, < 5 MIDP and at least 30 advanced minimally invasive gastrointestinal resections.

Outcome of patients who underwent either distal pancreatectomy by the consultant or registrars were compared.

Our primary outcome was the conversion rate. The secondary outcomes were 90-days postoperative outcomes including CR-POPF defined and classified according to the 2016 ISGPF definition.

ELIGIBILITY:
Inclusion criteria:

- Patients who underwent minimally invasive distale pancreatectomy for benign or borderline pathology between 2009-2020

Exclusion criteria:

* open distal pancreatectomy
* minimally invasive distal pancreatectomy for pancreatic cancer
* 20 first consecutive patients operated on by the consultant (learning curve)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent minimally invasive distale pancreatectomy for benign or borderline pathology
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
open conversion rate | 1 day
  Necessity to swith from minimally invasive approach to open approach during laparoscopy

SECONDARY OUTCOMES:
Duration of surgery | 1 day
  Duration of surgery
Intraoperative bloodloss | 1 day
  Intraoperative bloodloss
Intraoperative transfusion | 1 day
  Intraoperative transfusion
severe complications Clavien Dindo>3 | 90 days postoperative
  severe complications Clavien Dindo>3
postoperative complications | 90 days postoperative
  postoperative complications
clinically relevant postoperative fistula | 90 days postoperative
  clinically relevant postoperative fistula (2016 ISGPF definition)
lenght of hospital stay | 90 days postoperative
  lenght of hospital stay
readmission rate | 90 days postoperative
  readmission rate
reoperation rate | 90 days postoperative
  reoperation rate

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC